CLINICAL TRIAL: NCT02735525
Title: Feasibility Trial for Postoperative Wound Surveillance Using Smartphones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-1581
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Surgical Wound Infection
Keywords: telemedicine; smartphone
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone monitoring (Experimental): Intervention arm
  Interventions: Device: Smartphone monitoring

INTERVENTIONS:
Device: Smartphone monitoring — Patients will be trained to use the smartphone and the wound surveillance app prior to discharge. Patients will use the app from home to take send digital images of their postoperative wounds and answer a short survey, all of which will be transmitted to a secure database maintained by the UW Department of Surgery and accessible only to UW-employed study personnel. These data will be evaluated by one of three vascular surgery service nurse practitioners (NPs) daily. Patients who have concerning findings either in their images or in their survey answers will be contacted for further evaluation.

SUMMARY:
The proposed trial is a pilot to test a smartphone application (app) that will ultimately allow patients to take and transmit photos of their postoperative wounds from home and relay other symptom information. This protocol covers the single-institution pilot study of the app's use in the period between hospital discharge and a patient's first follow-up clinic visit. The investigators will recruit vascular surgery patients either preoperatively in clinic or in the post-operative, pre-discharge period following surgery to participate in the pilot. Using a training protocol refined in the usability-testing phase of the project, patients will be trained to use the smartphone and the wound surveillance app prior to discharge. Patients will use the app from home to take send digital images of their postoperative wounds and answer a short survey, all of which will be transmitted to a secure database maintained by the University of Wisconsin (UW) Department of Surgery and accessible only to UW-employed study personnel. These data will be evaluated by one of three vascular surgery service nurse practitioners (NPs) daily and entered into the medical record. Patients who have concerning findings either in their images or in their survey answers will be contacted for further evaluation. Smartphones will be provided to patients who do not have one of their own, through a partnership with AT&T. Sociodemographic and comorbidity data collected from the medical record will be kept at UW Department of Surgery on a secure server and accessible only to UW employed study personnel.

DETAILED DESCRIPTION:
Study duration: 3 years

Population Description:

Patients are typically older adults with multiple comorbid conditions and low health literacy. Caregivers may have a similar profile or may be younger with some technological experience (adult son or daughter).

Recruitment and Consent Screening for eligibility: On the outpatient side, study personnel will identify eligible participants from the vascular surgery clinic schedule. On the inpatient side, study personnel will identify eligible participants from the service inpatients with the assistance of service NPs and residents. Eligible patients will be approached by study personnel and the operating surgeon or service NP to discuss the project and obtain consent.

Enrollment/baseline: Research personnel will introduce the study, obtain consent, and perform the training to teach a patient or caregiver how to take a picture of a wound.

A written consent will be obtained after a thorough discussion of the study. All of this information will be explained in a non-technical fashion. Time will be provided to answer patient and caregiver questions or concerns about the study. Patients and caregivers will also be warned about the risks of a breach in confidentiality, and what measures will be taken to try and prevent this, and also what will be done in the instance it may happen.

Study Activities Subject identification and recruitment: Study personnel with clinical access will identify eligible participants from the medical record.

Data elements to be collected from the medical record following consent: age, sex, type of surgery, date of surgery, surgical complications, zip code (to determine rural/urban status and 4G coverage), and comorbidities (particularly cognitive impairment and motor functioning impairment).

Treatment/intervention period: Regardless of where patients have been recruited and consented, the patient and/or their caregiver will be trained to use the app in the post-operative, predischarge period; additional training will be provided on how to use the device, as necessary. Notes will be taken to document the success of training and to identify any potential areas for improvement in the training protocol. The study personnel will then explain the protocol for when the patient is discharged home and answer any questions the patient and/or their caregiver may have. Participants will be provided with an iPhone 5, which will be theirs to keep following study completion. Prior to assigning a smartphone to a participant, study personnel will be guided through a process to reset the device and erase any information that was stored on it from the prior user. Participants' names and medical record numbers are encrypted and stored only in the backend app and are never placed on the device.

When the patient is discharged from the hospital, they will then be asked to take a photograph of their surgical wound and answer a short survey about their wound and their general recovery using the smartphone app. This information will be transmitted via encrypted connection to a secure research server in the UW Department of Surgery. A composite screen will be created that displays all of the transmitted images as well as the responses to the survey questions within the app. Each afternoon, a service NP or study personnel with MD surgical training will review the data transmitted and complete a short form documenting the appearance of the surgical wound. Within the review screen, the reviewer can mark the data as already reviewed, which will move the record to an archive list. This form will be scanned into the patient's medical record if there is new evidence of a burgeoning complication; the image will remain on the department server and not be associated with the medical record. Any concerning findings will prompt a phone call from the surgical service nurse practitioner (NP) to the patient to gather more information and recommend additional intervention/treatment as indicated, which may include antibiotics or a clinic visit; upon detection of a burgeoning complication, usual care clinical protocol takes over (as if the patient had called with the concern). Additionally, contact information for the vascular surgery clinic and study personnel is provided at 2 points through the app itself, so that patients and their caregivers can easily call with questions or concerns.

If a patient has not submitted information in the past 24 hours, a study personnel will call the patient to discuss the protocol and any difficulties they may be having with completing it. The phone call will not be punitive, but will be aimed at decreasing study attrition, identifying reasons why patients are not compliant with the stated protocol, and identifying possible measures to improve the protocol. Three attempts will be made to contact an individual patient. All patients will receive a call 5-6 days following discharge to assess use of the app regardless of attrition status.

Specific Aims/Study Objectives:

Goal: Evaluate the effectiveness and feasibility of a protocol for post-discharge wound monitoring using a smartphone app and its ability to detect postoperative wound complications and reduce hospital readmissions in a vascular surgery patient population..

Hypotheses being tested:

H 1: With a well-designed app and training module, patients will be empowered by the opportunity to participate in their postoperative care and prevent potentially life threatening wound complications.

H 2: Through the use of this smartphone app in the post-discharge period, wound complications will be detected earlier than they would be otherwise and that the need for hospital readmissions will decrease.

Device Information App description: Screen shots uploaded as supplementary content. No information or photo is retained on the phone. UW Department of Surgery IT, the entity who developed the app, has ensured that the app is HIPAA-compliant. Neither photos generated in this study nor associated information will be stored directly to the phone's camera role.

Device specifications, packaging, labeling: Smartphones will be iPhone 5s or 6 purchased through collaboration with AT&T.

1. Device iOS devices running iOS 8 or higher. A pass code will be used to secure and encrypt the device.

Devices will be maintained using the Apple Profile Manager which will allow remote-wiping of devices, preventing the install of additional apps, and limiting of other device features.

The Wound App (mobile application) will be installed through the Apple Profile Manager. The Wound app will not save any protected health information into permanent storage on the device. Photos and responses will be held in application memory before being submitted back to a Department of Surgery web server.

If the user is idle for more than 10 minutes the app will time out.

Photos and responses will be released from memory after they have been submitted or after the app has timed out.

ELIGIBILITY:
Inclusion Criteria:

* Vascular surgery patient capable of independently completing protocol or who has an identifiable competent caregiver
* Incision >3 cm in length

Exclusion Criteria:

* No decisional capacity and absence of competent caregiver
* Identifying mark in area of the wound that would be capture in digital image of the wound
* Under age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Protocol completion | Assessed at 2 weeks from enrollment of each participant
  The percentage of participants who completed the app for the full length of the protocol (from the day of discharge to the day of scheduled clinic follow-up) without requiring a reminder phone call.

SECONDARY OUTCOMES:
Patient willingness to participate | Assessed at consent/enrollment of eligible patients
  The percentage of eligible patients approached to participate in the protocol, compared to the number who consent to participate.
Participant satisfaction | Assessed at 2 weeks from enrollment for each participant
  Participant surveys at the end of the protocol to determine satisfaction with the protocol and to identify areas for improvement.
Wound complication detection | Assessed daily through 2 weeks from enrollment for each participant
  Percentage of participants who received a phone call for a worrisome image or survey response.
Time needed to successfully complete the training module | Assessed at enrollment for each participant
  Number of minutes taken to train the patient/caregiver to complete the training including questions and teach-back. Goal: 30 min.
Burden of protocol on clinical workflow | Through study completion, an average of 6 months
  Total additional time required by NP to complete all their responsibilities for response review, averaged by patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Kent, MD, Principal Investigator — University of Wisconsin, Department of Surgery
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunter RL, Fernandes-Taylor S, Rahman S, Awoyinka L, Bennett KM, Weber SM, Greenberg CC, Kent KC. Feasibility of an Image-Based Mobile Health Protocol for Postoperative Wound Monitoring. J Am Coll Surg. 2018 Mar;226(3):277-286. doi: 10.1016/j.jamcollsurg.2017.12.013. Epub 2018 Jan 19. PMID 29366555
- [Derived] Fernandes-Taylor S, Gunter RL, Bennett KM, Awoyinka L, Rahman S, Greenberg CC, Kent KC. Feasibility of Implementing a Patient-Centered Postoperative Wound Monitoring Program Using Smartphone Images: A Pilot Protocol. JMIR Res Protoc. 2017 Feb 22;6(2):e26. doi: 10.2196/resprot.6819. PMID 28228369